CLINICAL TRIAL: NCT04285398
Title: Natural History Study of Retinitis Pigmentosa Due to RHO, PDE6a or PDE6b Mutations
Brief Title: Prospective Natural History Study of Retinitis Pigmentosa
Acronym: PHENOROD2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SparingVision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PHENOROD2
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Retinitis Pigmentosa
Keywords: RHO; PDE6A; PDE6B; Pathogenic Mutation; Prospective; Natural History; Retinal Disease; Eye Disease; Blindness; Inherited Eye Disease; Vision Disorder; Inherited Retinal Disorder; Rod-Cone Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Diseases; Eye Diseases; Blindness; Vision Disorders; Cone-Rod Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group 1 (Other): Four years follow up of patients with ophthalmic examination.
  Interventions: Other: Ophthalmic examinations
- Study Group 2 (Other): Four years follow-up of patients with ophthalmic examination and mobility testing.
  Interventions: Other: Ophthalmic examinations; Other: Mobility Test

INTERVENTIONS:
Other: Ophthalmic examinations — Slit-lamp examination, IntraOcular Pressure, Visual Acuity, Visual Field, Full-field Stimulus Threshold, Dark adaptometry, Color Vision testing, Optical Coherence Tomography, Fundus AutoFluorescence and Adaptive Optics imaging.
Other: Mobility Test — Functional test to evaluate mobility and postural condition of patients
  Arms: Study Group 2

SUMMARY:
This is natural history study of rods and cones degenerations in patients with Retinitis Pigmentosa (RP) caused by pathogenic mutations in RHO, PDE6a or PDE6b gene mutations.

DETAILED DESCRIPTION:
This is an open, longitudinal, prospective, multicentric study to describe the disease progression in patients with retinitis pigmentosa due to mutation in genes with selective expression in rods: rhodopsin (RHO), phosphodiesterase 6a (PDE6a) or phosphodiesterase 6b (PDE6b).RHO,PDE6A or PDE6B mutation.

ELIGIBILITY:
Inclusion Criteria:

* RP with mutations affecting the RHO, PDE6A and PDE6B genes
* Visual acuity ≥ 20/200 for at least one eye at inclusion visit
* Binocular Visual field diameter ≥ 5° as measured on the Goldmann III-4e isopter at inclusion visit
* Patients having signed the informed consent form
* Sufficient knowledge of the local language to ensure understanding of the tasks to be performed and the instructions received
* Patient affiliated to a Health Security System if they are included in a clinical site based in France (per law)

Exclusion Criteria:

* Patients with any other gene mutation known to be involved in RP
* Patients with other ocular disorder likely to impact the retinal function
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Spectral Domain Optical Coherence tomography (SD-OCT) | 1 year
  Progression of disease over time as measured by SD-OCT (EZ length, ELM length, ONL thickness, macular volume).
Fundus Autofluorescence (FAF) | 1 year
  Progression of disease as measured by FAF (Hyperautofluorescent ring)

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Progression of disease over time as measured by best corrected visual acuity (BCVA) (ETDRS, Snellen) and refraction
Visual field | 1 year
  Progression of disease over time as measured by kinetic and static visual fields
Full-field stimulus threshold (FST) | 1 year
  Progression of disease over time as measured by FST
Color vision | 1 year
  15 Hue Desaturated Lanthony
Dark adaptometry (DA) | 1 year
  Progression of disease over time as measured by DA

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Audo, MD, PhD, Principal Investigator — CHNO XV-XX Paris - CIC 1423
Locations (2):
- UPMC Eye Center, Pittsburgh, Pennsylvania, United States
- CHNO XV-XX Paris - CIC 1423, Paris, France